CLINICAL TRIAL: NCT02092493
Title: The Effect of Magnetic Endoscopic Imaging (ScopeGuide) on the Mental Workload of Endoscopists During Colonoscopy
Brief Title: The Effect of ScopeGuide on the Mental Workload of Endoscopist
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MEI1
Record Dates: First submitted 2014-03-12; First posted 2014-03-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Any Symptoms Requiring Colonoscopy
Keywords: ScopeGuide; Colonoscopy; Mental workload

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-ScopeGuide (No Intervention): This arm will have patients undertaking the procedure without ScopeGuide. All outcome measures will be recorded as usual
- ScopeGuide (Experimental): Patients have their colonoscopy done with ScopeGuide
  Interventions: Device: ScopeGuide

INTERVENTIONS:
Device: ScopeGuide — These patient will have their procedure undertake with the use of ScopeGuide, which provides a 3d configuration of the colonoscope in the patient
  Other Names: Magnetic endoscopic imaging
  Arms: ScopeGuide

SUMMARY:
ScopeGuide (Magnetic endoscopic imaging) is a device used during some colonoscopies which provides real-time 3D image of the shape and configuration of the colonoscope as it travels through the colon. Whilst it is being used in clinical practice in most units in the UK, it is not a device which is routinely used on all lists, and most departments do not own enough ScopeGuides to have on all lists. Studies have shown it can potentially aid colonoscopy by improving completion rates and times as well as patient comfort in selected endoscopists (persons who perform the colonoscopy). However data on its benefit have been conflicting.

Subjective mental workload (the individuals mental resources required as a result of the multiple demands placed on him/her from a task)in healthcare employees is known to be important for the performance and safety of healthcare delivery. Increased workload during task performance may increase fatigue, facilitate errors and lead to overall inferior performance.

In colonoscopy high mental workload could potentially be responsible for longer procedural time, lack of trainee learning, inadvertent missing of lesions in the bowel as well as poor technique leading to patient discomfort. The effect of the endoscopist mental workload on their performance and potential facilitators to reduce mental workload is an area that has been neglected in this field.

This study aims to look at the mental workload of endoscopist during colonoscopy and the effect ScopeGuide may have on this workload.

Hypothesis: The use of ScopeGuide during colonoscopy will reduce the mental workload of the endoscopist performing the procedure

ELIGIBILITY:
Inclusion Criteria:

* All endoscopist performing colonoscopy at University hospital Southampton endoscopy unit
* All adult patients attending diagnostic colonoscopy

Exclusion Criteria:

* Endoscopist preference
* Patients unable to give informed consent
* Patient preference
* Patients with new diagnosis of colonic cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
mental workload scores for endoscopist performing colonoscopy (represented by the NASA-task load index scores on a visual analogue scale (VAS) ranging from 0-600) | within 1 hour of beginning procedure
  This will be a brief VAS scale questionnaire carried out when the endoscopist reaches the caecum
Caecal intubation times, recorded in minutes and seconds | within 1 hour of beginning procedure
  this would be the time it takes from the beginning of the procedure to reaching the caecum

SECONDARY OUTCOMES:
Withdrawal time measured in minutes and second | within 1 hour of beginning procedure
Overall procedure times in minutes and seconds | within 1 hour of beginning procedure
-'Timing' of procedures (day & am/pm & order on list) | upto 1 hour before beginning procedure
Polyp detection | within 1 hour of beginning procedure
Patient comfort scores on a visual analogue scale | within 1 hour of completing procedure
Sedation dose measured in milligrams and micrograms | within 1 hour of completing procedure
Patient pre-endoscopy anxiety levels measured on visual analogue scale | upto 1 hour before beginning procedure

CONTACTS AND LOCATIONS:
Overall Officials: Imdadur Rahman, MBChB MRCP, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- University Hospital Southampton, Southampton, Hamshire, United Kingdom